CLINICAL TRIAL: NCT06041971
Title: Safety and Feasibility Testing of a Fully Closed Loop System in Adolescents and Adults with Higher Baseline HbA1c Values
Brief Title: Fully Closed Loop At Home (FCL@Home)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Virginia (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-1684
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Treatment Groups Randomized Crossover: Participants will be randomized 1:1 within each age cohort to either conduct the two-week control period before use of the AIDANET system (group A) or after use of the AIDANET system (group B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental): Two-week control period before the use of the AIDANET system.
  Interventions: Device: AIDANET system
- Group B (Experimental): Two-week control period after the use of the AIDANET system.
  Interventions: Device: AIDANET system

INTERVENTIONS:
Device: AIDANET system — The study will involve testing a new AID system designed to enable full closed loop control and consisting of the following elements: the diabetes assistant (DiAs) prototyping platform (MAF 2019), connected to a Tandem t:AP research insulin pump and a Dexcom G6 CGM, and implementing the University of Virginia (UVA) AIDANET algorithm.

SUMMARY:
Protocol Overview/Synopsis This study will be conducted at 3 sites, with each site performing a session with up to 6 participants with a lower HbA1c (<8.0%) in one of 3 age categories (26-60, 18-25, or 14-17 years) followed by a session of up to 6 additional participants with a higher HbA1c (8.0-12.0%) with the same age categories (26-60, 18-25, or 14-17 years). The trial will aim to complete a total of 36 participants: 12 total participants within each age category and 18 participants within each HbA1c category; 12 participants at each site. The study may enroll up to 70 participants to account for dropouts across the study. The study will be performed for 5 days and 4 nights at a local hotel/rental. Following the hotel session, participants will undergo a 7 day/6-night remote monitored at-home use session. The study will also conduct a two-week control period gathering data on glycemic control and insulin administration with the participants usual care therapy. Participants will be randomized 1:1, stratified by age cohort, to either group A (control period prior to AIDANET use) or group B (control period after AIDANET use).

ELIGIBILITY:
Inclusion Criteria:

1. Age either 14-17, 18-25, or 26-60 years at time of consent.
2. Clinical diagnosis of T1D, based on investigator assessment, of at least 1 year duration.
3. HbA1c either <8.0 or 8.0-12.0% at time of consent.
4. Currently using insulin for at least 6 months.
5. Willingness to follow the protocol and sign the informed consent (and assent as applicable).
6. Living with one or more parent/guardian or supportive companions knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.
7. For females, not currently known to be pregnant or breastfeeding.
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to switch to use a commercially approved personal insulin (e.g., lispro or aspart, or biosimilar approved products) within the study pump as directed by the study team.
10. Currently using an insulin pump for at least the prior 6 months. Any commercially approved pump, either open loop or hybrid closed loop may be used.
11. Willingness to suspend use of any personal CGM other than Dexcom G6 once the DiAs system is in use. Participants may use their own Dexcom G6 during the study period.
12. Willingness to use the study FCL system (CGM, pump, and phone) during the relevant study period.
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
14. Willingness to participate in all study procedures including the house/hotel session, exercise challenges (e.g., one hour per day during hotel), and to consume approximately 3 unannounced meals per day during the relevant portion of the supervised hotel session.
15. Access to internet at home and willingness to upload data during the study as needed.
16. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
17. Participant is proficient in reading and writing English.

Exclusion Criteria:

1. Plans to start a new non-insulin glucose-lowering agent (e.g., GLP-1 receptor agonists, Symlin, DPP-4 inhibitors, sulfonylureas). Participants may be on a stable dose of such an agent for at least the past month.
2. Current use of an SGLT-2 or SGLT-1/2 inhibitor due to risk of euglycemic DKA.
3. Hemophilia or any other bleeding disorder.
4. History of severe hypoglycemic event with seizure or loss of consciousness in the last 12 months.
5. History of DKA event in the last 12 months.
6. History of chronic renal disease (CKD3b or 4) or currently on peritoneal or hemodialysis.
7. History of adrenal insufficiency.
8. Currently being treated for a seizure disorder.
9. Hypothyroidism or hyperthyroidism that is not adequately treated.
10. Coronary artery disease or other heart condition that would prevent participation in moderate intensity exercise.
11. Use of oral or injectable steroids at the time of enrollment or within the last 4 weeks.
12. Planned surgery during the study period.
13. Known ongoing adhesive intolerance that is not well managed.
14. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk.
15. Participation in another interventional trial at the time of enrollment.
16. Participant does not have a direct supervisor involved in the conduct of the trial.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Mean Sensor Glucose Value | Change between second week of the control period and the one-week at home period
  The primary metric for analysis will be change in mean sensor glucose value between the second week of the control usual-care period and the one-week remote monitored at-home FCL period.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Forlenza, MD, Principal Investigator — University of Colorado Anschutz - Barbara Davis Center
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Barbara Davis Center, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No